CLINICAL TRIAL: NCT00678535
Title: Open-label, Randomized, Controlled, Multicenter Phase III Study Investigating Cetuximab in Combination With Capecitabine (Xeloda, X) and Cisplatin (P) Versus XP Alone as First-line Treatment for Subjects With Advanced Gastric Adenocarcinoma Including Adenocarcinoma of the Gastroesophageal Junction
Brief Title: Erbitux in Combination With Xeloda and Cisplatin in Advanced Esophago-gastric Cancer
Acronym: EXPAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200048-052; 2007-004219-75 (EudraCT Number)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Gastric Cancer
Keywords: 1st line treatment for Gastric Cancer; Cetuximab; Capecitabine; Xeloda; Cisplatin; Progression-free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab plus Capecitabine plus Cisplatin (Experimental)
  Interventions: Drug: Cetuximab; Drug: Capecitabine; Drug: Cisplatin
- Capecitabine plus Cisplatin (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Cetuximab — Single first dose of cetuximab 400 milligram per square meter (mg/m^2) will be administered intravenously over 120 minutes followed by weekly intravenous infusion of cetuximab 250 mg/m^2 over 60 minutes in each 3-week treatment cycle, until documented disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: Erbitux
  Arms: Cetuximab plus Capecitabine plus Cisplatin
Drug: Capecitabine — Capecitabine 1000 mg/m^2 will be administered orally twice daily from evening of Day 1 to morning of Day 15 for every 3-week treatment cycle, until documented disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: Xeloda
Drug: Cisplatin — Cisplatin 80 mg/m^2 will be administered intravenously with infusion over 1 to 4 hours on Day 1 of each 3-week treatment cycle, until documented disease progression, unacceptable toxicity, or withdrawal of consent.

SUMMARY:
The primary objective of this study is to demonstrate that addition of cetuximab to 1st-line treatment with capecitabine (Xeloda, X) and cisplatin (P) [XP] chemotherapy regimen has a clinically relevant benefit for subjects with advanced gastric adenocarcinoma including gastroesophageal junction (GEJ) adenocarcinoma, in terms of progression free survival (PFS).

Secondary objectives are to assess cetuximab plus XP versus XP alone with respect to overall survival, overall tumor response, quality of life (QoL) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before any study-related activities are carried out
* Age greater than or equal to (>=) 18 years
* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (Adenocarcinoma of the gastroesophageal junction [AEG] Types I-III according to Siewert classification)
* Archived tumor material sample for at least subsequent standardized Epidermal Growth Factor Receptor (EGFR) expression assessment
* Unresectable advanced (M0) or unresectable metastatic (M1) disease
* At least one radiographically documented measurable lesion in a previously non-irradiated area according to response evaluation criteria in solid tumors (RECIST). The primary tumor site is to be considered as a non-measurable lesion only
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Estimated life expectancy greater than (>) 12 weeks
* Medically accepted contraception (if the risk of conception exists)
* Glomerular filtration rate (GFR) >= 60 milliliter per minute (mL/min) The GFR is based on the Cockcroft-Gault formula for creatinine clearance
* Aspartate-aminotransferase (ASAT) less than or equal to (=<) 2.5 * upper limit of normal (ULN) and alanine-aminotransferase (ALAT) =< 2.5 *ULN
* Bilirubin =< 3 * ULN
* Absolute neutrophil count (ANC) >= 1.5 * 10^9 per liter
* Platelets >= 100 * 10^9 per liter
* Hemoglobin >=10 gram per deciliter (g/dL) (without transfusions)
* Sodium and potassium within normal limits or =< 10 percent above or below (supplementation permitted)

Exclusion Criteria:

* Prior chemotherapy, however, previous (neo-)adjuvant (radio-) chemotherapy allowed if finished > 1 year prior to start of study treatment and no more than 300 mg/m^2 cisplatin has been administered
* Prior treatment with an antibody or molecule targeting EGFR and/or Vascular Endothelial Growth Factor Receptor (VEGFR) related signaling pathways
* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Radiotherapy (except localized radiotherapy for pain relief), major surgery or any investigational drug within 30 days before the start of study treatment
* Concurrent chronic systemic immune or hormone therapy not indicated in this study protocol (except for physiologic replacement)
* Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the 12 months before study Screening, or high risk of uncontrolled arrhythmia
* Active Hepatitis B or C
* Chronic diarrhea or short bowel syndrome
* Presence of any contra-indication to treatment with cetuximab, capecitabine and cisplatin including:

  * Known hypersensitivity to capecitabine, fluorouracil, cisplatin, cetuximab or to any of the excipients of these drugs
  * Known dihydropyrimidine dehydrogenase (DPD) deficiency
  * Hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
  * Current treatment with sorivudine or chemically related analogues, such as brivudine
  * Symptomatic peripheral neuropathy National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade >= 2 and/or ototoxicity NCI CTCAE Grade >= 2, except if due to trauma or mechanical impairment due to tumor mass
* Pregnancy or lactation period
* Concurrent treatment with a non-permitted drug
* Treatment in another clinical study within 30 days prior to study screening
* Previous malignancy other than gastric cancer within 5 years prior to study screening, except for basal cell cancer of the skin or pre-invasive cancer of the cervix
* Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
* Legal incapacity or limited legal capacity
* Significant disease which, in the Investigator's opinion, would exclude the subject from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, MD, PhD, Principal Investigator — University Clinic Leipzig, University Cancer Center Leipzig (UCCL), Leipzig Germany
Locations (130):
- Research site, Rosario, Argentina
- Australia (3):
  - Research site, Coburg VIC
  - Research site, Frankston, VIC
  - Research site, Perth
- Austria (5):
  - Research site, Graz
  - Research site, Kufstein
  - Research site, Steyr
  - Research Site, Vienna
  - Research Site, Zams
- Belgium (3):
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research site, Verviers
- Brazil (7):
  - Research site, Campinas
  - Research site, Ijuí
  - Research site, Jaú
  - Research site, Porto Alegre
  - Research site, Salvador
  - Research site, Santo André
  - Research site, Sâo Paulo
- Bulgaria (4):
  - Research site, Pleven
  - Research site, Plovdiv
  - Research site, Rousse
  - Research site, Sofia
- Chile (4):
  - Research site, Reñaca
  - Research site, Santiago
  - Research site, Temuco
  - Research site, Valparaíso
- China (6):
  - Research site, Beijing
  - Research site, Guangzhou
  - Research site, Hefei
  - Research site, Nanjing
  - Research site, Shanghai
  - Research site, Shenyang
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research site, Prague
- France (6):
  - Research site, Besançon
  - Research site, Clermont-Ferrand
  - Research site, La Roche-sur-Yon
  - Research site, Marseille
  - Research site, Paris
  - Research site, Rennes
- Germany (24):
  - Research Site, Berlin
  - Research site, Bielefeld
  - Research site, Braunschweig
  - Research site, Cologne
  - Research Site, Dresden
  - Research Site, Essen
  - Research site, Esslingen am Neckar
  - Research site, Frankfurt
  - Research Site, Giessen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research site, Ludwigshafen
  - Research Site, Mainz
  - Research Site, München
  - Research site, Offenbach
  - Research Site, Regensburg
  - Research Site, Schwäbisch Hall
  - Research site, Schweinfurt
  - Research site, Stuttgart
  - Research Site, Timisoara
  - Research Site, Troisdorf
  - Research site, Ulm
  - Research site, Weiden
  - Research Site, Weilheim
- Greece (2):
  - Research site, Ioannina
  - Research site, Thessaloniki
- Research site, Hong Kong, Hong Kong
- Hungary (4):
  - Research site, Budapest
  - Research site, Győr
  - Research Site, Kaposvár
  - Research Site, Tatabánya
- Israel (5):
  - Research site, Haifa
  - Research site, Jerusalem
  - Research site, Petach Tiqva
  - Research site, Ramat Gan
  - Research site, Tel Aviv
- Italy (6):
  - Research site, Ancona
  - Research site, Bologna
  - Research site, Milan
  - Research site, Napoli
  - Research site, Roma
  - Research site, Rozzano (Milano)
- Japan (11):
  - Research site, Chiba
  - Research site, Ehime
  - Research site, Hokkaido
  - Research site, Kōtoku
  - Research site, Nagoya
  - Research site, Osaka
  - Research site, Saitama
  - Research site, Shizuoka
  - Research site, Tochigi
  - Research site, Tokyo
  - Research site, Yokohama
- Poland (4):
  - Research site, Gdansk
  - Research site, Lublin
  - Research site, Opole
  - Research site, Wroclaw
- Research site, Sana Maria Da Feira, Portugal
- Romania (5):
  - Research site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research site, Timișoara
- Russia (4):
  - Research site, Kazan'
  - Research site, Moscow
  - Research site, Obninsk
  - Research site, Saint Petersburg
- South Korea (5):
  - Research site, Anyang
  - Research site, Daegu
  - Research site, Inchon-si
  - Research site, Seongnam
  - Research Site, Seoul
- Spain (7):
  - Research Site, Alicante
  - Research site, El Palmar-Murcia
  - Research site, Lugo
  - Research site, Pamplona
  - Research Site, Santander
  - Research site, Seville
  - Research Site, Valencia
- Taiwan (7):
  - Research site, Changhua
  - Research site, Kaohsiung City
  - Research site, Kaohsiung County
  - Research site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research site, Taoyuan District
- United Kingdom (2):
  - Research site, Guildford
  - Research site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): June 2008/December 2010. Clinical data cut-off: 31 March 2012 Study completion 17 February 2013.
Pre-assignment Details: Enrolled: 1,191 screened for eligibility; 287 excluded (mainly non-fulfillment of inclusion or exclusion criteria). 904 participants randomized.
Groups:
- Cetuximab Plus Capecitabine Plus Cisplatin: Cetuximab weekly (initial dose 400 milligram per square meter [mg/m^2] followed by 250 mg/m^2 intravenous infusion), cisplatin (3-week cycle, 80 mg/m^2 intravenous infusion on Day 1) and capecitabine (3-week cycle, 1000 mg/m^2 orally twice daily for 14 days ) until documented disease progression, unacceptable toxicity, or withdrawal of consent.
- Capecitabine Plus Cisplatin: Cisplatin (3-week cycle, 80 mg/m^2 intravenous infusion on Day 1) and capecitabine (3-week cycle, 1000 mg/m^2 orally twice daily for 14 days) until documented disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Started | 455 (ITT population) | 449 (ITT population)
Completed | 362 (subjects who died before or at 31 March 2012) | 351 (subjects who died before or at 31 March 2012)
Not Completed | 93 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin | Total
Number analyzed (Participants) | 455 | 449 | 904
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.16) | 58.5 (10.83) | 58.3 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 231
  Male | 339 | 334 | 673

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time: Independent Review Committee (IRC) Assessments
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause within 60 days of the last tumor assessment or randomization. Participants without event are censored on the date of last tumor assessment.
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, 30 Jun 2008 until cut-off date (31 Mar 2012)
Population: Intent-to-treat (ITT) population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 455 | 449
months | 4.4 [4.2 to 5.5] | 5.6 [5.1 to 5.7]
Statistical Analysis 1: Comparison: Cetuximab Plus Capecitabine Plus Cisplatin vs Capecitabine Plus Cisplatin; Primary efficacy analysis: To test equality of progression free survival time between treatment groups, applying the two-sided stratified log-rank test (randomization strata: disease stage, previous oesophagectomy/gastrectomy and prior(neo-) adjuvant(radio) chemotherapy, α=5%); Test type: Superiority or Other; p = 0.3158, Stratified log rank; Hazard Ratio (HR) = 1.091, 95% CI [0.920 to 1.292] — Kaplan-Meier method was used to estimate median PFS time. HR was calculated using Cox proportional hazards model stratified by randomization strata

2. Secondary Outcome: Overall Survival (OS)
Description: The OS time is defined as the time from randomization to death or last day known to be alive. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, that is, 30 Jun 2008 until cut-off date, (31 Mar 2012)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 455 | 449
months | 9.4 [8.3 to 10.6] | 10.7 [9.4 to 11.3]
Statistical Analysis 1: Comparison: Cetuximab Plus Capecitabine Plus Cisplatin vs Capecitabine Plus Cisplatin; To test equality of OS time between treatment groups, applying the two-sided stratified log-rank test (randomization strata: disease stage, previous oesophagectomy/gastrectomy and prior (neo-) adjuvant(radio) chemotherapy, α=5%); Test type: Superiority or Other; p = 0.9547, Stratified log rank; Hazard Ratio (HR) = 1.004, 95% CI [0.866 to 1.165] — Kaplan-Meier method was used to estimate median OS time. HR was calculated using Cox proportional hazards model stratified by randomization strata

3. Secondary Outcome: Best Overall Response (BOR) Rate: Independent Review Committee (IRC) Assessments
Description: The BOR rate is defined as the percentage of participants having achieved complete response (CR) or partial response (PR) as the best overall response, based on radiological assessments (based on response evaluation criteria in solid tumors [RECIST] Version 1.0) from the IRC.
Time Frame: Every 6 weeks until progression, reported between day of first participant randomized, that is, 30 Jun 2008 until cut-off date, (31 Mar 2012)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 455 | 449
percentage of participants | 29.9 [25.7 to 34.3] | 29.2 [25.0 to 33.6]
Statistical Analysis 1: Comparison: Cetuximab Plus Capecitabine Plus Cisplatin vs Capecitabine Plus Cisplatin; The best overall response rate was compared with the Cochran-Mantel-Haenszel test (strata: disease stage, previous oesophagectomy/gastrectomy and prior(neo-) adjuvant(radio) chemotherapy, two-sided with α=5%); Test type: Superiority or Other; p = 0.7696, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.0435, 95% CI [0.7844 to 1.3882]

4. Secondary Outcome: Quality of Life (QoL) Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: Mean global health status and social functioning scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a better QoL.
Time Frame: Baseline, Week 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60, reported between day of first participant randomized, that is, 30 Jun 2008 until cut-off date (31 Mar 2012)
Population: Analysis population included participants who had at least one evaluable EORTC QLQ-C30 questionnaire and were also included in the ITT population. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 450 | 430
units on a scale
  Global health status: Baseline | 57.49 (22.168) | 57.19 (22.124)
  Global health status: Week 6 | 59.00 (21.879) | 61.80 (22.089)
  Global health status: Week 12 | 60.17 (20.796) | 63.35 (22.077)
  Global health status: Week 18 | 60.45 (20.015) | 61.83 (21.499)
  Global health status: Week 24 | 62.46 (22.978) | 63.61 (19.477)
  Global health status: Week 30 | 63.65 (21.722) | 64.11 (19.757)
  Global health status: Week 36 | 65.06 (22.629) | 57.72 (21.602)
  Global health status: Week 42 | 59.29 (21.558) | 62.64 (22.005)
  Global health status: Week 48 | 63.39 (21.317) | 66.67 (19.395)
  Global health status: Week 54 | 60.63 (16.198) | 66.67 (14.651)
  Global health status: Week 60 | 62.50 (13.918) | 61.81 (17.210)
  Social functioning status: Baseline | 74.36 (27.077) | 76.52 (26.601)
  Social functioning status: Week 6 | 68.94 (28.885) | 75.70 (27.415)
  Social functioning status: Week 12 | 71.48 (26.547) | 75.65 (27.691)
  Social functioning status: Week 18 | 71.22 (25.317) | 75.51 (25.612)
  Social functioning status: Week 24 | 74.20 (26.143) | 78.26 (27.633)
  Social functioning status: Week 30 | 78.51 (24.766) | 76.67 (24.962)
  Social functioning status: Week 36 | 76.28 (21.730) | 73.58 (22.353)
  Social functioning status: Week 42 | 68.57 (27.348) | 78.16 (22.318)
  Social functioning status at Week 48 | 80.36 (22.705) | 78.00 (23.432)
  Social functioning status: Week 54 | 74.71 (27.682) | 80.56 (27.371)
  Social functioning status: Week 60 | 78.33 (23.632) | 68.06 (32.144)

5. Secondary Outcome: Quality of Life (QoL) Assessed by EuroQol 5Dimensions (EQ-5D) Questionnaire
Description: EQ-5D questionnaire is a measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 single items are combined to obtain a single index score that is health utility index (HUI) score reflecting subject's preferences for different health states. The lowest possible score is -0.59 and the highest is 1.00, higher scores on the EQ-5D represent a better QoL.
Time Frame: as for outcome 4
Population: Analysis population included participants who had at least one evaluable EuroQoL EQ-5D questionnaire and were also included in the ITT population. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 450 | 430
units on a scale
  Baseline | 0.743 (0.240) | 0.749 (0.235)
  Week 6 | 0.739 (0.276) | 0.769 (0.254)
  Week 12 | 0.752 (0.239) | 0.775 (0.246)
  Week 18 | 0.742 (0.251) | 0.755 (0.235)
  Week 24 | 0.733 (0.300) | 0.761 (0.265)
  Week 30 | 0.737 (0.301) | 0.790 (0.230)
  Week 36 | 0.710 (0.311) | 0.711 (0.309)
  Week 42 | 0.722 (0.209) | 0.689 (0.307)
  Week 48 | 0.719 (0.227) | 0.770 (0.216)
  Week 54 | 0.733 (0.275) | 0.730 (0.191)
  Week 60 | 0.760 (0.322) | 0.742 (0.170)

6. Secondary Outcome: Safety - Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Time from first dose up to Day 30 after last dose of study treatment, reported between day of first participant randomized, that is, 30 Jun 2008 until cut-off date (31 Mar 2012)
Population: The safety population included all participants who received at least one dose of any trial treatment that is, cetuximab, cisplatin, or capecitabine.
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Number analyzed (Participants) | 446 | 436
participants | 446 | 432

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment.
Description: An AE is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Cetuximab Plus Capecitabine Plus Cisplatin | Capecitabine Plus Cisplatin
Serious Adverse Events (participants affected / at risk) | 239/446 | 194/436
Other Adverse Events (participants affected / at risk) | 441/446 | 429/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Capecitabine Plus Cisplatin (N=446) | Capecitabine Plus Cisplatin (N=436)
Anaemia (Blood and lymphatic system disorders) | 10 | 17
Neutropenia (Blood and lymphatic system disorders) | 9 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 3 | 1
Myocardial infarction (Cardiac disorders) | 3 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 4
Myocardial ischaemia (Cardiac disorders) | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Auricular perichondritis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 16 | 25
Diarrhoea (Gastrointestinal disorders) | 15 | 15
Nausea (Gastrointestinal disorders) | 11 | 13
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Ascites (Gastrointestinal disorders) | 9 | 3
Dysphagia (Gastrointestinal disorders) | 6 | 3
Ileus (Gastrointestinal disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Obstruction gastric (Gastrointestinal disorders) | 3 | 2
Subileus (Gastrointestinal disorders) | 3 | 1
Melaena (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 5
Gastric perforation (Gastrointestinal disorders) | 1 | 1
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 12 | 13
Fatigue (General disorders) | 11 | 5
Pyrexia (General disorders) | 8 | 7
Disease progression (General disorders) | 7 | 1
Asthenia (General disorders) | 6 | 5
Mucosal inflammation (General disorders) | 3 | 3
Performance status decreased (General disorders) | 3 | 3
Device dislocation (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 0
Device occlusion (General disorders) | 1 | 0
Stent malfunction (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Death (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 0 | 4
Pain (General disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 1
Bile duct stenosis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 4 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Sepsis (Infections and infestations) | 5 | 2
Pneumonia (Infections and infestations) | 4 | 8
Device related infection (Infections and infestations) | 3 | 4
Gastroenteritis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 3 | 0
Paronychia (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 5
Blood urine (Investigations) | 1 | 0
Electrocardiogram low voltage (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Troponin I increased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 15 | 3
Dehydration (Metabolism and nutrition disorders) | 9 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 9
Hypophagia (Metabolism and nutrition disorders) | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 6 | 4
Cerebral infarction (Nervous system disorders) | 5 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 3 | 4
Renal failure acute (Renal and urinary disorders) | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 26 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 11 | 2
Hypotension (Vascular disorders) | 2 | 2
Peripheral ischaemia (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 2
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Capecitabine Plus Cisplatin (N=446) | Capecitabine Plus Cisplatin (N=436)
Neutropenia (Blood and lymphatic system disorders) | 194 | 234
Anaemia (Blood and lymphatic system disorders) | 127 | 155
Thrombocytopenia (Blood and lymphatic system disorders) | 81 | 89
Leukopenia (Blood and lymphatic system disorders) | 67 | 94
Tinnitus (Ear and labyrinth disorders) | 20 | 23
Nausea (Gastrointestinal disorders) | 273 | 265
Diarrhoea (Gastrointestinal disorders) | 172 | 105
Vomiting (Gastrointestinal disorders) | 165 | 192
Constipation (Gastrointestinal disorders) | 120 | 110
Stomatitis (Gastrointestinal disorders) | 100 | 41
Abdominal pain (Gastrointestinal disorders) | 92 | 72
Abdominal pain upper (Gastrointestinal disorders) | 67 | 44
Dyspepsia (Gastrointestinal disorders) | 45 | 21
Dysphagia (Gastrointestinal disorders) | 23 | 14
Fatigue (General disorders) | 187 | 162
Asthenia (General disorders) | 92 | 98
Mucosal inflammation (General disorders) | 65 | 31
Pyrexia (General disorders) | 64 | 38
Oedema peripheral (General disorders) | 27 | 26
Hyperbilirubinaemia (Hepatobiliary disorders) | 25 | 11
Paronychia (Infections and infestations) | 63 | 3
Weight decreased (Investigations) | 107 | 77
Haemoglobin decreased (Investigations) | 37 | 37
Glomerular filtration rate decreased (Investigations) | 30 | 35
Blood creatinine increased (Investigations) | 29 | 37
Aspartate aminotransferase increased (Investigations) | 26 | 13
Alanine aminotransferase increased (Investigations) | 24 | 16
Neutrophil count decreased (Investigations) | 20 | 22
Platelet count decreased (Investigations) | 17 | 22
Decreased appetite (Metabolism and nutrition disorders) | 221 | 201
Hypomagnesaemia (Metabolism and nutrition disorders) | 133 | 60
Hypokalaemia (Metabolism and nutrition disorders) | 86 | 56
Hypocalcaemia (Metabolism and nutrition disorders) | 67 | 38
Hyponatraemia (Metabolism and nutrition disorders) | 42 | 34
Hypoalbuminaemia (Metabolism and nutrition disorders) | 39 | 24
Dehydration (Metabolism and nutrition disorders) | 29 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 29 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 19
Dizziness (Nervous system disorders) | 66 | 45
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 27
Dysgeusia (Nervous system disorders) | 32 | 29
Headache (Nervous system disorders) | 31 | 22
Neuropathy peripheral (Nervous system disorders) | 23 | 41
Paraesthesia (Nervous system disorders) | 20 | 27
Insomnia (Psychiatric disorders) | 41 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 21
Hiccups (Respiratory, thoracic and mediastinal disorders) | 29 | 47
Rash (Skin and subcutaneous tissue disorders) | 194 | 23
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 162 | 97
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 78 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 56 | 11
Acne (Skin and subcutaneous tissue disorders) | 54 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 19
Skin fissures (Skin and subcutaneous tissue disorders) | 28 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 15 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other